CLINICAL TRIAL: NCT01392313
Title: Measurement of Glomerular Filtration Rate (GFR) Using Iohexol in Healthy Subjects Taking Creatinine Supplements
Brief Title: Measurement of Renal Function With Iohexol in Subjects Ingesting Carnitine
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 10-03-068
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Carnitine Ingestion
Keywords: carnitine, kidney
MeSH Terms: interventions — Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: Yes

ARMS (2):
- Carnitine (Experimental): Participants will be given Creatinine supplements
  Interventions: Dietary Supplement: Carnitine
- Placebo (Placebo Comparator): participants will be given creatinine placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Carnitine — Carnitine Ingestion
  Arms: Carnitine
Dietary Supplement: Placebo — Carnitine placebo
  Arms: Placebo

SUMMARY:
The investigators will measure renal function in subjects ingesting carnitine to determine if the product alters renal function.

ELIGIBILITY:
Inclusion Criteria:

* carnitine ingestion

Exclusion Criteria:

* renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Iohexol clearance | 1 month
  Iohexol clearance will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Joel Neugarten, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States